CLINICAL TRIAL: NCT06312748
Title: Novel Approaches for Improving Vascular Function in Veterans With HFpEF
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Collaborators: University of Utah (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: CARB-019-20S; 138675 (Other: University of Utah)
Record Dates: First submitted 2024-03-08; First posted 2024-03-15 (Actual); Last update posted 2025-06-19 (Actual); Status verified 2025-06

CONDITIONS: Heart Failure With Preserved Ejection Fraction; Inflammation
Keywords: vascular health; exercise tolerance; HFpEF; nitric oxide
MeSH Terms: conditions — Inflammation | interventions — Citrulline; sapropterin; Atorvastatin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: A block randomization method will be used to randomize participants into equal groups and will be handled by investigational pharmacist.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (6):
- L-Citrulline, Then Placebo (Experimental): Participants will receive a 90-day supply of L-Citrulline and perform baseline assessments of resting arterial blood pressure, ECT, arterial elasticity/pulse contour analysis, flow-mediated vasodilation and passive limb movement procedures. Participants will return to the laboratory for up to 5 additional study visits (days 10, 20, 30, 60, and 90) and repeat the experimental protocol. After a two-week washout period, participants will receive a 90-day supply of Placebo and perform baseline and follow-up assessments as above.
  Interventions: Drug: L-Citrulline; Drug: Placebo for L-Citrulline
- BH4, Then Placebo (Experimental): Participants will receive a 90-day supply of BH4 and perform baseline assessments of resting arterial blood pressure, ECT, arterial elasticity/pulse contour analysis, flow-mediated vasodilation and passive limb movement procedures. Participants will return to the laboratory for up to 5 additional study visits (days 10, 20, 30, 60, and 90) and repeat the experimental protocol. After a two-week washout period, participants will receive a 90-day supply of Placebo and perform baseline and follow-up assessments as above.
  Interventions: Drug: BH4; Drug: Placebo for BH4
- Atorvastatin, Then Placebo (Experimental): Participants will receive a 90-day supply of Atorvastatin and perform baseline assessments of resting arterial blood pressure, ECT, arterial elasticity/pulse contour analysis, flow-mediated vasodilation and passive limb movement procedures. Participants will return to the laboratory for up to 5 additional study visits (days 10, 20, 30, 60, and 90) and repeat the experimental protocol. After a two-week washout period, participants will receive a 90-day supply of Placebo and perform baseline and follow-up assessments as above.
  Interventions: Drug: Atorvastatin; Drug: Placebo for Atorvastatin
- Placebo, Then L-Citrulline (Experimental): Participants will receive a 90-day supply of Placebo and perform baseline assessments of resting arterial blood pressure, ECT, arterial elasticity/pulse contour analysis, flow-mediated vasodilation and passive limb movement procedures. Participants will return to the laboratory for up to 5 additional study visits (days 10, 20, 30, 60, and 90) and repeat the experimental protocol. After a two-week washout period, participants will receive a 90-day supply of L-Citrulline and perform baseline and follow-up assessments as above.
  Interventions: Drug: L-Citrulline; Drug: Placebo for L-Citrulline
- Placebo, Then BH4 (Experimental): Participants will receive a 90-day supply of Placebo and perform baseline assessments of resting arterial blood pressure, ECT, arterial elasticity/pulse contour analysis, flow-mediated vasodilation and passive limb movement procedures. Participants will return to the laboratory for up to 5 additional study visits (days 10, 20, 30, 60, and 90) and repeat the experimental protocol. After a two-week washout period, participants will receive a 90-day supply of BH4 and perform baseline and follow-up assessments as above.
  Interventions: Drug: BH4; Drug: Placebo for BH4
- Placebo, Then Atorvastatin (Experimental): Participants will receive a 90-day supply of Placebo and perform baseline assessments of resting arterial blood pressure, ECT, arterial elasticity/pulse contour analysis, flow-mediated vasodilation and passive limb movement procedures. Participants will return to the laboratory for up to 5 additional study visits (days 10, 20, 30, 60, and 90) and repeat the experimental protocol. After a two-week washout period, participants will receive a 90-day supply of Atorvastatin and perform baseline and follow-up assessments as above.
  Interventions: Drug: Atorvastatin; Drug: Placebo for Atorvastatin

INTERVENTIONS:
Drug: L-Citrulline — 100 mg tablet
  Arms: L-Citrulline, Then Placebo; Placebo, Then L-Citrulline
Drug: Placebo for L-Citrulline — L-Citrulline-matched Placebo tablet
  Arms: L-Citrulline, Then Placebo; Placebo, Then L-Citrulline
Drug: BH4 — 10mg/kg
  Other Names: Kuvan®, sapropterin dihydrochloride
  Arms: BH4, Then Placebo; Placebo, Then BH4
Drug: Placebo for BH4 — BH4-matched Placebo
  Arms: BH4, Then Placebo; Placebo, Then BH4
Drug: Atorvastatin — 10 mg tablet
  Other Names: Lipitor®
  Arms: Atorvastatin, Then Placebo; Placebo, Then Atorvastatin
Drug: Placebo for Atorvastatin — Atorvastatin-matched Placebo
  Arms: Atorvastatin, Then Placebo; Placebo, Then Atorvastatin

SUMMARY:
This project will evaluate the impact of L-Citrulline, tetrahydrobiopterin (BH4), and atorvastatin administration on physical capacity and vascular function in Veterans with heart failure with preserved ejection fraction (HFpEF).

DETAILED DESCRIPTION:
The hospital admission rate for Veterans with heart failure with a preserved ejection fraction (HFpEF) continues to rise within the VA Health Care System, making HF the number one reason for hospital discharge Additionally, readmission rates of Veterans with HF tend to be higher than the national average, emphasizing the shortcomings of current therapeutic strategies Indeed, while optimized pharmacotherapy has led to a declining mortality in heart failure with reduced ejection fraction (HFrEF) patients, similar therapies in patients with HFpEF have been unsuccessful in altering the natural history of the disease Clearly, alternative therapeutic approaches are needed to improve outcomes in this ever-growing Veteran patient group.

The clinical presentation of HFpEF continues to be defined by dyspnea upon exertion and severe exercise intolerance symptoms that are unlikely due to a simple deficit in cardiac mechanics Indeed, the contribution of vascular dysfunction to exercise intolerance in patients with HFpEF has recently been identified highlighting the importance of disease-related changes in the peripheral circulation to HFpEG pathophysiology. While the mechanisms responsible for vascular dysfunction in HFpEF have not been established, there is an emerging concept that chronic inflammation and the associated production of reactive oxygen species (ROS), stemming from HFpEF-associated comorbidities and inactivity, plays a crucial role. The proposed work seeks to address this important knowledge gap by examining the mechanisms linking inflammation, vascular health, and exercise tolerance in Veterans with HFpEF, and identifying which aspects of this cascade could be targeted to improve outcomes in this patient group.

In HFpEF, the peripheral vasculature represents an area that is particularly vulnerable to the harmful effects of circulating ROS due to the interaction with nitric oxide (NO). Indeed, following formation and release from the endothelium, the fate of NO is dictated to a large degree by the presence of ROS that catalyze the formation of peroxynitrite (ONOO-), thereby decreasing NO bioavailability. This deleterious effect on NO formation is amplified by ONOO--mediated oxidation of tetrahydrobiopterin (BH4), effectively "uncoupling" endothelial nitric oxide synthase (eNOS) and thus further diminishing NO production. Bioavailability of NO may also be diminished through reductions in precursor (L-Arginine/L-Citrulline) availability, such that a "substrate limitation" may also be present in patients with HFpEF.

While the potential of increased NO bioavailability to improve outcomes in patients with HFpEF has been increasingly recognized, results from clinical trials utilizing NO donors have been largely negative, suggesting a more comprehensive approach may be needed. Thus, the overall goal of the project is to evaluate the mechanisms responsible for vascular dysfunction and exercise intolerance in Veterans with HFpEF, which will be accomplished through selective pharmacologic targeting of distinct pathways known to regulate vascular NO signaling. The investigators have identified three discreet points in the cascade from inflammation to vascular dysfunction that may represent therapeutic targets for improving exercise tolerance in patients with HFpEF, and thus propose a series of integrative aims that will combine novel methodology with targeted pharmacologic interventions to selectively determine the importance of NO substrate, enzymatic cofactor bioavailability, and statin-induced mitigation of inflammation and ROS to disease-related changes in inflammation and NO signaling in HFpEF.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older and able to give written informed consent.
* New York Heart Association (NYHA) functional class I, II, or III.
* Left Ventricular Ejection Fraction (LVEF) > 50%.
* Plasma Brain Natriuretic Peptide (BNP) equal to or greater than 150 pg/mL or NT-proBNP equal to or greater than 600 pg/mL at Visit 1, or a BNP equal to or great than 100 pg/mL (or NT-proBNP equal to or greater than 400 pg/mL) and a hospitalization for heart failure within the last 12 months.

Exclusion Criteria:

* History of hypersensitivity or allergy to any lipophilic statin.
* Prior EF <50%.
* NYHA Class IV.
* Patients with HFpEF secondary to significant uncorrected primary valvular disease.
* Active liver disease or unexplained persistent elevations in serum transaminase.
* Women who are pregnant or may become pregnant.
* Patients currently treated with antioxidants, nitrates, PDE-5 inhibitors, or statins.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2021-05-19 (Actual); Primary Completion 2028-09-30 (Estimated); Study Completion 2030-09-30 (Estimated)

PRIMARY OUTCOMES:
Flow-mediated dilation (FMD) | Baseline, Day 90
  Peak change in brachial artery diameter (%)

SECONDARY OUTCOMES:
Passive Limb Movement (PLM) | Baseline, Day 90
  Peak change in leg blood flow (ml/min)

CONTACTS AND LOCATIONS:
Overall Officials: David W. Wray, PhD, Principal Investigator — VA Salt Lake City Health Care System, Salt Lake City, UT
Locations (1):
- VA Salt Lake City Health Care System, Salt Lake City, UT, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: No